CLINICAL TRIAL: NCT06379217
Title: A Phase I, Open-label, Multi-center Exploratory Safety and Efficacy Study With PSMA, SSTR2 and GRPR Targeted Radioligand Therapy in Metastatic Neuroendocrine Prostate Cancer.
Brief Title: NEPC Study: An Exploratory Safety and Efficacy Study With PSMA, SSTR2 and GRPR Targeted Radioligand Therapy in Metastatic Neuroendocrine Prostate Cancer.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617H12101; 2023-505655-43 (EudraCT Number)
Record Dates: First submitted 2024-03-04; First posted 2024-04-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Neuroendocrine Prostate Cancer
Keywords: [68Ga]Ga-PSMA-11; [177Lu]Lu-PSMA-617; [68Ga]Ga-DOTA-TATE; [177Lu]Lu-DOTA-TATE; [68Ga]Ga-NeoB; [177Lu]Lu-NeoB; Neuroendocrine prostate cancer (NEPC); Metastatic Neuroendocrine Prostate Cancer (mNEPC); Radioligand Imaging (RLI); Radioligand Therapy (RLT); Prostate-specific membrane antigen (PSMA); Somatostatin Receptor 2 (SSTR2); Gastrin Releasing Peptide Receptor (GRPR); Phase 1
MeSH Terms: interventions — gallium 68 PSMA-11; gallium Ga 68 dotatate; Gallium; Lutetium; Lutetium-177; copper dotatate CU-64; Gonadotropin-Releasing Hormone; Antiemetics; Metoclopramide

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a treatment arm based on their predominantly expressed target per PET images (based on central read):
  * [177Lu]Lu-PSMA-617 will be assigned to those with predominant PSMA expression
  * [177Lu]Lu-DOTA-TATE will be assigned to those with predominant SSTR2 expression
  * [177Lu]Lu-NeoB will be assigned to those with predominant GRPR expression
  In complex cases the local Investigator has the authority to make decisions on the most appropriate RLT assignment.
  If the selected RLT assignment is to a treatment arm that has reached its maximum enrollment, the patient will not be able to receive the selected RLT and will not join the treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PSMA-predominant NEPC (Experimental)
  Interventions: Drug: [68Ga]Ga-PSMA-11; Drug: [68Ga]GA-DOTA-TATE; Drug: [68Ga]Ga-NeoB; Drug: [177Lu]Lu-PSMA-617; Drug: Gonadotropin-releasing hormone (GnRH) analogues; Drug: GnRH antagonists
- SSTR2-predominant NEPC (Experimental)
  Interventions: Drug: [68Ga]Ga-PSMA-11; Drug: [68Ga]GA-DOTA-TATE; Drug: [68Ga]Ga-NeoB; Drug: [177Lu]Lu-DOTA-TATE; Drug: L-Lysine HCl-L-Arginine HCl, 2.5 %,; Drug: Gonadotropin-releasing hormone (GnRH) analogues; Drug: GnRH antagonists; Drug: Antiemetics & antinauseants; Drug: Metoclopramide
- GRPR-predominant NEPC (Experimental)
  Interventions: Drug: [68Ga]Ga-PSMA-11; Drug: [68Ga]GA-DOTA-TATE; Drug: [68Ga]Ga-NeoB; Drug: [177Lu]Lu-NeoB; Drug: Gonadotropin-releasing hormone (GnRH) analogues; Drug: GnRH antagonists

INTERVENTIONS:
Drug: [68Ga]Ga-PSMA-11 — [68Ga]Ga-PSMA-11 will be administered as a single intravenous dose of approximately 150 MBq (4 mCi) to be administered during baseline imaging and at any time ≥ 6 weeks after first RLT dose. Sites should consider doing PET/CT imaging with RLT corresponding RLI as the first of three PET/CT scans. Administered dose should not be lower than 111 MBq (3 mCi) or higher than 259 MBq (7 mCi)
  Other Names: Gallium (68Ga) gozetotide
Drug: [68Ga]GA-DOTA-TATE — [68Ga]Ga-DOTA-TATE will be administered as a single intravenous dose to be administered during baseline imaging and at any time ≥ 6 weeks after first RLT dose. Sites should consider doing PET/CT imaging with RLT corresponding RLI as the first of three PET/CT scans. within a range of 100-200MBq (2.7-5.4 mCi)
  Other Names: Gallium (68Ga) DOTA-TATE
Drug: [68Ga]Ga-NeoB — [68Ga]Ga-NeoB will be administered as a single intravenous dose to be administered during baseline imaging and at any time ≥ 6 weeks after first RLT dose. Sites should consider doing PET/CT imaging with RLT corresponding RLI as the first of three PET/CT scans. within a range of 150-250 MBq (4.1-6.8 mCi).
  Other Names: Gallium (68Ga) NeoB
Drug: [177Lu]Lu-PSMA-617 — [177Lu]Lu-PSMA-617 will be administered as an intravenous infusion at a dose of 7.4 GBq (200mCi) (+/- 10%), every 6 weeks for 6 cycles.
  Other Names: Lutetium (177Lu) vipivotide tetraxetan
  Arms: PSMA-predominant NEPC
Drug: [177Lu]Lu-DOTA-TATE — [177Lu]Lu-DOTA-TATE will be administered as an intravenous infusion at a dose of 7.4 GBq (200mCi) (+/- 10%) every 6 weeks for 6 cycles.
  Other Names: Lutetium (177Lu) DOTA-TATE
  Arms: SSTR2-predominant NEPC
Drug: [177Lu]Lu-NeoB — [177Lu]Lu-NeoB will be administered as an intravenous infusion at a dose of 9.25 GBq (250mCi) every 6 weeks for 6 cycles
  Other Names: Lutetium (177Lu) NeoB
  Arms: GRPR-predominant NEPC
Drug: L-Lysine HCl-L-Arginine HCl, 2.5 %, — sterile solution for infusion Lysine HCl-Arginine HCl, 2.5 % (1L)
  Other Names: Lysine HCl-Arginine HCl, 2.5 %
  Arms: SSTR2-predominant NEPC
Drug: Gonadotropin-releasing hormone (GnRH) analogues — Anatomical Therapeutic Chemical [ATC] code L02AE
Drug: GnRH antagonists — abarelix, degarelix, or relugolix
Drug: Antiemetics & antinauseants — ATC code A04A
  Arms: SSTR2-predominant NEPC
Drug: Metoclopramide — ATC code A03FA01
  Arms: SSTR2-predominant NEPC

SUMMARY:
The purpose of this study is to evaluate the change in the expression of treatment targets on the surface of tumor cells (Prostate Specific Membrane Antigen (PSMA), Somatostatin Receptor 2 (SSTR2), and Gastrin Releasing Peptide Receptor (GRPR) between the baseline and following targeted radioligand therapy (RLT). Study will use radioligand imaging (RLI) to determine predominantly expressed target on the surface of tumor cells. Based on predominant expression of target, corresponding RLT targeting PSMA, SSTR2, or GRPR RLT will be given for up to 6 cycles every 6 weeks as intravenous (i.v.) injection in participants with metastatic neuroendocrine prostate cancer (mNEPC).

Study is planning to enroll approximately 20 participants in [177Lu]Lu-PSMA-617 treatment arm, approximately 3 participants in [177Lu]Lu-NeoB treatment arm, and approximately 13 participants in [177Lu]Lu-DOTA-TATE treatment arm.

DETAILED DESCRIPTION:
The screening period for each participant includes imaging with 3 radioligand imaging (RLI) compounds to assess expression level of PSMA, SSTR2 and GRPR. Participants will be assigned to the radioligand treatment (RLT) corresponding to their predominantly expressed target based on blinded independent central review (BICR). During the treatment period, participants will receive up to 6 cycles of the assigned RLT, corresponding to a total dose of 44.4 GBq (+/-10%) for [177Lu]Lu-PSMA-617 or [177Lu]Lu-DOTA-TATE , and 55.5 GBq (+/-10%) for [177Lu]Lu-NeoB. No crossover to a different type of RLT is allowed.

At least six weeks after receiving the first cycle of RLT, participants must be scanned again with up to 3 RLIs but must be scanned, with at least with one RLI corresponding to the received RLT, which is recommended to be performed first. All post-baseline PET/CT scans should be performed using the same PET/CT imaging agent and same PET/CT camera, acquisition and reconstruction protocols as used for screening PET/CT for the participant.

The post-treatment follow-up period consists of a 42-days post EOT safety follow-up visit, efficacy, and survival follow-up until radiographic disease progression, death, lost to follow-up or withdrawal of consent, whichever occurs first.

The planned duration of treatment is up to 36 weeks for all treatment arms in this study, with treatment given every 6 weeks ±7 days. Participants may be discontinued from treatment earlier due to unacceptable toxicity or disease progression, and/or at the discretion of the Investigator or the participant.

ELIGIBILITY:
Key Inclusion criteria:

* Participants must have metastatic prostate cancer with neuroendocrine differentiation as determined by at least one of the following:

  1. Histologically small cell or neuroendocrine cancer from a primary prostate or metastatic biopsy confirmed by local laboratory.
  2. Expression of NEPC markers (e.g., chromogranin or synaptophysin) in tumor tissue by IHC confirmed by local laboratory
  3. Progression of visceral metastases in the absence of PSA progression
  4. Serum chromogranin A > 5x normal limit, or neuron-specific enolase > 2x normal limit with control for proton-pump inhibitors (PPI) drugs among concomitant treatment
  5. Prostate adenocarcinoma with molecular features of neuroendocrine differentiated cancer (e.g., 2 of the following 3: PTEN, TP53, or RB loss)
* PSMA and/or SSTR2 and/or GRPR PET-positive participants, with at least one measurable lesion per RECIST 1.1 with moderate target expression in at least one of the 3 PET/CT scans per BICR assessment
* Castrate level of serum/plasma testosterone (< 50 ng/dl, or < 1.7 nmol/L) for participants with adenocarcinoma component or stable testosterone level for participants with pure neuroendocrine carcinoma
* Recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapy
* Participant has adequate bone marrow and organ function (as assessed by central laboratory for eligibility)
* ECOG status =< 2

Key Exclusion criteria:

* Previous treatment with any of the following within 6 months prior to Screening: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation
* Previous PSMA, SSTR2, or GRPR targeted radioligand therapy
* Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy or investigational therapy
* History of CNS metastases that are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for study participants

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must have metastatic prostate cancer
Enrollment: 28 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Number/extent of lesions with at least a moderate uptake of any of the Radioligand Imaging (RLI) | Baseline (baseline imaging is performed during the 42 day screening period)
  Number/extent of lesions with at least a moderate update of any of the RLIs according to visual assessment scoring scale on each corresponding targeted PET/CT scan based on blinded independent central review (BICR) assessment.
Percentage changes in quantitative PET parameters. | Post-Baseline (from date of baseline imaging scans to post-baseline scans, at least 6 weeks after receiving the first cycle of radioligand treatment)
  Percentage changes in quantitative PET/CT parameters (SUVmax, SUVmean, SUVpeak, target-positive Tumor Volume (target -TV), Total Lesion (target (TL-target)] and changes in number of target-positive lesions (as per visual assessment) on each corresponding target PET/CT based on BICR.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From date of assignment to one of the treatment arms until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 31 months
  Overall Response Rate (ORR) is defined as the proportion of participants with the best overall response (BOR) of confirmed complete response (CR) or partial response (PR) based on Prostate Cancer Working Group 3 (PCWG3) modified-RECIST v1.1.
Disease Control Rate (DCR) | From date of assignment to one of the treatment arms until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 31 months
  Disease Control Rate (DCR) is defined as the proportion of participants with BOR of CR, PR, stable disease (SD), or non-CR/non-PD based on PCWG3 modified-RECIST v1.1.
Duration of response (DOR) | From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to approximately 31 months
  Duration of response (DOR) is defined as the time (in months) from the date of the first confirmed response (CR or PR) to the date of first documented progression according to PCWG3 modified-RECIST v1.1 or death due to any cause, among participants with a confirmed response.
Radiographic Progression-free Survival (rPFS) | From date of assignment to one of the treatment arms until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 31 months
  Radiographic Progression-free Survival (rPFS) is defined as the time from the date of first dose of study treatment to the date of first documented radiographic progression (as assessed by the local investigator and using PCWG3 modified-RECIST v1.1 criteria) or death due to any cause.
Proportion of participants with a decline in PSA level | Baseline, Cycle 1 Day 1 (each cycle is 42 days), Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, End Of Treatment, 6 weeks after End of Treatment
  The PSA analysis will investigate the proportion of participants with a decline in PSA level from baseline to each visit.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) for Radioligand Therapy (RLT) | Up to 42 days after last dose administration (Safety Follow-up) and every 12 weeks until end of long term follow up (Long-term FU) for selected AEs and SAEs
  The distribution of adverse events for Radioligand Therapy (RLT) will be done via the analysis of frequencies for Adverse Events (AEs) and Serious Adverse Events (SAEs) through the monitoring of relevant clinical and laboratory safety parameters.
  Adverse event monitoring should be continued for at least 42 days following the end of treatment (EOT) visit.
  Participants receiving the study treatment [68Ga]Ga-DOTA-TATE/[177Lu]Lu-PSMA-617 or [177Lu]Lu-NeoB will continue to be followed for safety every 12 weeks during the long-term follow-up for selected adverse events.
Dose modifications for [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Up to 42 days after last dose administration (Safety Follow-up)
  Dose modifications (dose interruptions, dose discontinuations and reductions) for [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB will be assessed and summarized using descriptive statistics.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) for Radioligand Imaging (RLI) | Continuously from informed consent for the first 6 weeks and selected AEs and SAEs thereafter
  The distribution of adverse events for Radioligand Imaging (RLI) will be done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs) through the monitoring of relevant clinical and laboratory safety parameters.
Blood radioactivity concentration of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE, [177Lu]Lu-NeoB) | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs, 2 hrs, 4 hrs, 6 hrs 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Data will be listed by participant and visit/sampling time point. Descriptive summary statistics will be provided by visit/sampling time point and treatment arm including the frequency (n, %) of concentrations below the lower limit of quantification (LLOQ) and reported as zero.
Blood mass concentration of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE, [177Lu]Lu-NeoB) | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs, 2 hr, 4 hr, 6 hrs, 24 hrs, 48 hrs 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Data will be listed by participant and visit/sampling time point. Descriptive summary statistics will be provided by visit/sampling time point and treatment arm including the frequency (n, %) of concentrations below the lower limit of quantification (LLOQ) and reported as zero.
Observed maximum blood concentrations (Cmax) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs , 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Time of maximum blood concentration (Tmax) occurence of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hours (h), 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Area under the blood concentration time curve (AUC) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs , 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC will be listed and summarized using descriptive statistics.
Total systemic clerance (CL) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs, 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase (Vz) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs, 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Terminal half-life (T^1/2) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days) pre-dose, post-dose/end of infusion (EOI) and then 0.5 hrs, 2 hrs, 4 hrs, 6 hrs, 24 hrs, 48 hrs, 168 hrs post EOI. Cycle 3 Day 1 EOI, 1 hr, 48 hrs post EOI. Cycle 5 Day 1 EOI, and then 1 hr, 48 hrs post EOI.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-life will be listed and summarized using descriptive statistics.
Absorbed radiation doses of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days), Cycle 1 Day 2, Cycle 1 Day 3, Cycle 1 Day 8, Cycle 3 Day 1, Cycle 3 Day 3, Cycle 5 Day 1, Cycle 5 Day 3 (Cycle 3 Day 2, Cycle 3 Day 8, Cycle 5 Day 2 and Cycle 5 Day 8 where required by local authorities)
  The analysis of biodistribution and dosimetry endpoints will consist of descriptive summaries and graphical presentations of the derived parameters. For each of the treatments, the absorbed dose by body organs and tumor lesions will be determined by calculation of TACs obtained from the radiotracer uptake (as percentage of injected dose) in selected organs and lesions (coming from image quantification).
Time Activity Curves (TACs) of [177Lu]Lu-PSMA-617, [177Lu]Lu-DOTA-TATE and [177Lu]Lu-NeoB | Cycle 1 Day 1 (each cycle is 42 days), Cycle 1 Day 2, Cycle 1 Day 3, Cycle 1 Day 8, Cycle 3 Day 1, Cycle 3 Day 3, Cycle 5 Day 1, Cycle 5 Day 3 (Cycle 3 Day 2, Cycle 3 Day 8, Cycle 5 Day 2 and Cycle 5 Day 8 where required by local authorities)
  The analysis of biodistribution and dosimetry endpoints will consist of descriptive summaries and graphical presentations of the derived parameters. For each of the treatments, the absorbed dose by body organs and tumor lesions will be determined by calculation of TACs obtained from the radiotracer uptake (as percentage of injected dose) in selected organs and lesions (coming from image quantification).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (4):
  - Stanford University, Palo Alto, California
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Novartis Investigative Site, Nantes, France
- Germany (2):
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rostock
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: No